CLINICAL TRIAL: NCT02275403
Title: Randomised Clinical Trial of Acupuncture Plus Standard Care Versus Standard Care for Chemotherapy Induced Peripheral Neuropathy (CIPN)
Brief Title: Standard Care Alone or With Acupuncture for CIPN in Breast Cancer and Multiple Myeloma
Acronym: ACUFOCIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Emmie Taylor, Clinical Trials Project Manager, The Christie NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12_DOG06_165; PB-PG-0213-30129 (Other Grant/Funding Number: NIHR Research for Patient Benefit); CFTSp062 (Other: Sponsor)
Record Dates: First submitted 2014-10-22; First posted 2014-10-27 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Multiple Myeloma; Gastrointestinal Cancer; Gynaecological Cancer
MeSH Terms: conditions — Breast Neoplasms; Multiple Myeloma; Gastrointestinal Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Standard care plus acupuncture (Experimental): Medication taken to manage the symptom burden of CIPN plus acupuncture
  Interventions: Procedure: Acupuncture; Other: Medication taken to manage the symptom burden of CIPN
- Arm B: Standard care alone (Active Comparator): Medication taken to manage the symptom burden of CIPN
  Interventions: Other: Medication taken to manage the symptom burden of CIPN

INTERVENTIONS:
Procedure: Acupuncture — 10 x weekly sessions (40 minutes per session) of acupuncture by a trained therapist.
  Arms: Arm A: Standard care plus acupuncture
Other: Medication taken to manage the symptom burden of CIPN — Standard of care medication to manage CIPN symptoms, as determined by a clinician in accordance with local trust policy. The standard care for CIPN includes a variety of oral medications to manage the altered sensations caused by damage to the peripheral nerves. These oral medications include, but are not limited to; Gabapentin, Amitriptyline and Pregabalin. In addition, medicated creams and gels may be used.

SUMMARY:
The purpose of this study is to determine whether the addition of acupuncture to standard treatment reduces the level of chemotherapy induced peripheral neuropathy experienced by patients with breast cancer, multiple myeloma, gastrointestinal cancer or gynaecological cancer during or following treatment with neurotoxic chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy Induced Peripheral Neuropathy (CIPN) is a significant clinical challenge for patients receiving specific chemotherapy regimen (e.g. taxanes and Bortezomib) and critically, if severe, CIPN can lead to the discontinuation of life prolonging treatment. CIPN poses a major problem for patient care as standard pharmacological treatments for CIPN have been found to be commonly ineffective and are often inadequate due to dosing complexities, delayed analgesic onset and side effects.

A service evaluation of the clinical data secured from using acupuncture to manage CIPN symptoms over a period of 18 months at The Christie National Health Service (NHS) Foundation Trust suggests it has the potential to provide an efficacious management tool to be used in addition to standard medication. This aim of this trial is to formally evaluate a 10 week course of acupuncture in the management of CIPN of grade 2 or above (symptoms experienced have a functional impact, graded in accordance with CTCAE v4.03), in patients with breast cancer, multiple myeloma, gastrointestinal cancer or gynaecological cancer.

This is a randomised, phase II, single-centre, controlled, open label trial . Patients meeting eligibility criteria will be randomised to receive acupuncture plus standard care (treatment arm) or standard care alone (control arm). Patients in both arms of the study will receive standard medication to manage symptoms of CIPN, as determined by a clinician in accordance with local trust policy. In addition to this, patients randomised to the treatment arm will receive 40 minute sessions of acupuncture on a weekly basis for 10 weeks. All patients will be offered acupuncture, to commence off trial at the end of their 10 week study period.

Outcome measures have been focused on assessing the impact of acupuncture on the patients' quality of life, symptom burden of CIPN and quantifying any effect size. There will also be a preliminary health economic evaluation of cost effectiveness. The data will be disseminated in addition to being used to establish whether a larger, multisite trial to confirm efficacy across all diagnostic groups, user acceptability and cost effectiveness is appropriate. This work will facilitate the team validating the study protocol and design as a template for a multicentre study and confirm user acceptability of the approach through additional qualitative data collected through focus group work at the completion of study participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer, multiple myeloma, gastrointestinal cancer or gynaecological cancer who are receiving or who have received neurotoxic chemotherapy treatment for their condition
* The capacity to understand the patient information sheet and the ability to give written informed consent
* Willingness and ability to comply with scheduled visits and study procedures, including the self-report QoL questionnaires and patient diaries
* Age ≥ 18 years; no upper age limit
* CIPN of ≥ Grade II (CTCAE v4.03)
* Platelet count of ≥ 30 x 10*9/L
* Neutrophil count of ≥ 0.5 x 10*9/L
* MYMOP2 score of their most troubling CIPN symptom ≥ 3

Exclusion Criteria:

* Patients who have previously received acupuncture for neuropathy
* Patients who have received acupuncture for any indication, other than neuropathy, within the previous 6 months
* Women who are pregnant or breast feeding
* Co-morbidity with a bleeding disorder
* Patients with an aversion to needles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04-13 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Change in Measure Yourself Medical Outcome Profile (MYMOP2) score of the most troubling symptom of CIPN | Baseline, week 6 and week 10
  Assessed from patient completed questionnaire data: MYMOP2

SECONDARY OUTCOMES:
Change in grade of CIPN | Baseline, week 6 and week 10
  Assessed by a clinician using a set of standardised questions, as a prompt, to assess the functional impact of CIPN. CIPN will be graded in accordance with CTCAE v4.03
Change in use of concomitant CIPN related medication | Up to 10 weeks after baseline
  Includes change in dose and change in medication used to manage the symptom burden of CIPN.
Change in chemotherapy dosage | Up to 10 weeks after baseline
Pain related scores | Up to 10 weeks after baseline
  Captured by the patient at baseline and then daily in the patient diary from week 1
Quality of life | Baseline, week 6 and week 10
  Assessed from patient completed questionnaire data: European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) and the associated CIPN20 module
Acupuncture treatment compliance | From week 1 (start of acupuncture treatment) until week 10
  Compliance to attending weekly acupuncture sessions
Preliminary health economic evaluation of cost effectiveness | Up to 10 weeks after baseline
  Data will be captured from patient diaries completed continuously from week 1 until week 10 and from the patient notes. Patients will also complete the Euroqol (EQ-5D-5L) questionnaire at baseline, week 6 and week 10.
Uptake of the offer of acupuncture at 10 weeks | 10 weeks
  All patients will be offered acupuncture, to commence after the 10 week study period, at the 6 week visit. Acceptance of the offer will be captured at the 10 week visit.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wardley, Study Chair — The Christie NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Oldham Hospital, Oldham

IPD SHARING:
Plan to Share IPD: No